CLINICAL TRIAL: NCT00676845
Title: Effect of Olmesartan Medoxomil on Arterial Stiffness and Thickness in Subjects With Metabolic Syndrome
Brief Title: Study to Determine if Olmesartan Medoxomil Has the Potential to Benefit the Cardiovascular System in Terms of Arterial Protection
Acronym: ArtStiff
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo Europe, GmbH, a Daiichi Sankyo Company (Industry)
Responsible Party: Sponsor
Organization: Daiichi Sankyo (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DSE-866/47; 2007-003131-23 EudraCT number
Record Dates: First submitted 2008-05-08; First posted 2008-05-13 (Estimated); Last update posted 2018-12-24 (Actual); Status verified 2012-04

CONDITIONS: Metabolic Syndrome; Hypertension
Keywords: Arterial stiffness; Vascular protection
MeSH Terms: conditions — Metabolic Syndrome; Hypertension | interventions — Olmesartan Medoxomil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Placebo Comparator): A 3-week placebo run-in period.
  Interventions: Drug: placebo
- 2 (Experimental): Olmesartan medoxomil oral tablets, at lowest study dosage for 52-week double-blind treatment period
  Interventions: Drug: olmesartan medoxomil
- 3 (Experimental): Olmesartan medoxomil oral tablets at the lowest dosage for 4 weeks followed by a higher dosage for 48 weeks.
  Interventions: Drug: olmesartan medoxomil
- 4 (Experimental): Olmesartan medoxomil oral tablets at the lowest dosage for 4 weeks followed by a higher dosage for 4 weeks followed by the highest study dose for 44 weeks.
  Interventions: Drug: olmesartan medoxomil

INTERVENTIONS:
Drug: olmesartan medoxomil — dosage form: oral tablet; frequency: daily; duration: 52 weeks
  Arms: 2
Drug: placebo — dosage form: tablet; frequency: daily; duration: 3 weeks
  Arms: 1
Drug: olmesartan medoxomil — dosage form: oral tablet; frequency: daily; duration: 52 weeks
  Arms: 3
Drug: olmesartan medoxomil — dosage form: oral tablet; frequency: daily; duration: 52 weeks
  Arms: 4

SUMMARY:
This study will analyse the dose-dependent effect of olmesartan medoxomil on the change in arterial stiffness in subjects with hypertension and metabolic syndrome

ELIGIBILITY:
Inclusion Criteria:

* Male and female outpatients
* Age greater than or equal to 18 years and less than or equal to 75 years
* Hypertension and metabolic syndrome defined, according to the ATP III/IDF 2005 and ESH/ESC 2007 definitions, as BP greater than or equal to 130/85 mmHg and <150/95 mmHg (i.e. untreated high normal BP or "low range" mild hypertension) and at least 2 of the following traits at:
* Abdominal obesity (waist circumference >102 cm for men and >88 cm for women)
* Triglyceride level greater than or equal to 150 mg/dL
* High density lipoprotein (HDL) <40 mg/dL for men and <50 mg/dL for women
* Fasting blood glucose greater than or equal to 110 mg/dL and <126 mg/dL (i.e. no type 2 diabetes)
* No anti-hypertensive treatment or treatment with only one anti-hypertensive medication within the last 3 months. Note: treatment with angiotensin II receptor blockers (ARB)or angiotensin-converting enzyme inhibitors (ACE) is not allowed within the last 6 months.

Exclusion Criteria:

* Pregnant or lactating female (prerequisite for female subjects of childbearing potential: adequate contraception)
* Type 1 and type 2 diabetes
* "High range" mild hypertension (i.e. systolic blood pressure [SBP]: 150 - <160 mmHg and /or diastolic blood pressure [DBP]: 95 - <100 mmHg)
* Moderate (SBP: 160 - 179 mmHg and DBP: 100 - 109 mmHg), severe (SBP: greater than or equal to 180 mmHg and/or greater than or equal to 110 mmHg), or resistant (hypertension resistant to treatment)hypertension
* Secondary hypertension of any aetiology, such as renal disease, pheochromocytoma, or Cushing's syndrome

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2008-08; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
The change from baseline in carotid-femoral pulse wave velocity (PWV) | Up to 1 year of double-blind treatment
The change from baseline in carotid-femoral PWV, after adjustment for change from baseline in mean blood pressure (MBP)as measured at the same visit | Up to 1 year of double-blind treatment

SECONDARY OUTCOMES:
On blood pressure (BP) lowering, assessed by conventional BP measurement and 24h ambulatory BP measurement (24h-ABPM) | Up to 1 year of double-blind treatment
On central pulse pressure (PP) and augmentation index (AI) | Up to 1 year of double-blind treatment
On common carotid stiffness, intima-media thickness (IMT), and internal diameter | Up to 1 year of double-blind treatment

CONTACTS AND LOCATIONS:
Locations (3):
- Ghent, Belgium
- Nuremberg, Germany
- Monza, Italy

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Laurent S, Boutouyrie P; Vascular Mechanism Collaboration. Dose-dependent arterial destiffening and inward remodeling after olmesartan in hypertensives with metabolic syndrome. Hypertension. 2014 Oct;64(4):709-16. doi: 10.1161/HYPERTENSIONAHA.114.03282. Epub 2014 Jul 7. PMID 25001274